CLINICAL TRIAL: NCT05968716
Title: Addressing Unmet Social Needs Among Hospitalized Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 1K08HS028473-01A1 (AHRQ); 1K08HS028473-01A1 (AHRQ)
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Social Needs Screening; Caregiver-care Team Relationships; Social Needs Status; Child Health Status; Caregiver Health Status; Utilization, Health Care
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: The investigators will utilize a before-and-after trial design, whereby the "control group" consists of caregivers studied before a social needs screening protocol is implemented on a pediatric hospital ward, and the "intervention group" consists of caregivers studied after a social needs screening protocol is implemented on a pediatric hospital ward.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (pre-implementation) arm (No Intervention): Caregivers recruited from the pediatric hospital ward before the social needs screening and intervention protocol is implemented will compose the "control" group or pre-implementation group.
- Intervention (post-implementation) arm (Experimental): Caregivers recruited from the pediatric hospital ward after the social needs screening and intervention protocol is implemented will compose the "intervention" group or post-implementation group.
  Interventions: Other: Social needs screening protocol

INTERVENTIONS:
Other: Social needs screening protocol — Pediatric hospital ward stakeholders will develop and implement a social needs screening protocol designed to screen families of hospitalized children for social risk factors and then provide resources to address their social needs. The intervention will consist of the protocol that is developed and implemented.
  Arms: Intervention (post-implementation) arm

SUMMARY:
The purpose of this pilot study is to determine the feasibility and acceptability of implementing a social needs screening and intervention protocol in the pediatric inpatient setting by conducting a pilot trial on a pediatric ward. The investigators' hypothesis is that it will be feasible and acceptable to implement a social needs screening and intervention protocol. The investigators will work with pediatric word healthcare team members to develop a social needs screening and intervention protocol. They will then compare preliminary health and social outcome measures between children hospitalized during the pre-intervention period (control group) vs. the post-intervention period (intervention group).

DETAILED DESCRIPTION:
Millions of children in the US live in families with unmet social needs, and numbers increased during the COVID-19 pandemic. Children with unmet social needs are at increased risk of experiencing worse health and health care outcomes, and addressing unmet social needs can improve health and reduce health care utilization. Consequently, many professional organizations now endorse screening for and addressing social needs in clinical settings. However, despite social needs screening recommendations, there are no established best practices for clinical settings, and there has not been much focus on the pediatric inpatient setting. In order to understand whether identifying and addressing social needs in the pediatric inpatient setting positively impacts social and health outcomes, interventions must be developed and assessed that seek to accomplish this. Before launching large trials to assess such interventions, the feasibility and acceptability of implementing social needs interventions in the pediatric inpatient setting must determined. The objective of this pilot study is to determine the feasibility and acceptability of implementing a social needs screening and intervention protocol in the pediatric inpatient setting by conducting a pilot trial on a pediatric ward. The investigators' hypothesis is that it will be feasible and acceptable to implement a social needs screening and intervention protocol in this setting.

The investigators will utilize a before-and-after trial design to assess feasibility, acceptability, process, and preliminary outcome measures of implementing a social needs screening and intervention protocol in a tertiary children's hospital. Caregivers of hospitalized pediatric patients will be eligible to participate in surveys about screening acceptability and social and health outcomes if they are over 18 and their child is hospitalized on the transitional care general pediatrics unit within the 4 months prior to implementation of the protocol (control/pre-implementation group) or 4 months after the wash-in period (intervention/post-implementation group). Nurses, social workers, case managers, nurse practitioners, and physicians will be eligible to participate in a survey about protocol acceptability and satisfaction if they worked on the unit after protocol implementation.

A study team member will approach caregivers and ask if they would be potentially interested in filling out a survey about their experiences with being screened for social needs during their hospitalization and being contacted in 90 days for a follow-up survey. If interested, a study team member will screen the caregiver for eligibility and then obtain caregiver informed consent before administering the baseline survey. The consent will include a HIPAA authorization form to enable access to EHR records for the purposes of extracting utilization data (e.g., missed follow-up appointments). A follow-up survey will be administered via phone 3 months later. For care team members, an email will be sent to unit staff requesting participation in a voluntary survey regarding the social needs protocol with a link to the consent and survey included.

The investigators' goal is to recruit 25 caregivers in both the pre- and post-period, for a total of 50 caregivers. For the care team member survey, the hope is to gain as many members' input as possible. Based on the employee engagement response at the study site, the investigators believe that emailing roughly 93 care team members will respond.

The investigators will develop a social needs screening and intervention protocol for the ward based on: 1) input from unit leaders and stakeholders; 2) interviews from caregivers and care team members conducted previously. The goal is to develop and implement the protocol with a multidisciplinary group of unit stakeholders in 6 months.

Children hospitalized within the 4 months prior to intervention implementation will serve as the control group. Children hospitalized after a two-month "wash-in" period after protocol implementation will represent the intervention group. Post-intervention data will be collected for 4 months after implementation. The pilot will consist of roughly 50 caregivers of children and 93 care team members of the inpatient ward. This will allow us to estimate effect sizes for a future multi-site randomized clinical trial. Although The investigators may detect some intervention effects, the goal of the pilot is to assess feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver's child is hospitalized in the Transitional Care Unit (TCU) of Benioff Children's Hospital - San Francisco
* English or Spanish Speaking
* Parent/caregiver accompanying a patient hospitalized 0-17 years old
* Consenting adult over or equal to 18 years old
* Initially admitted to the TCU
* Caregiver's child is part of a service for which pediatric residents or advance practice providers provide care

Exclusion Criteria:

* Non-English or non-Spanish speaking caregiver
* Caregiver under age 18
* Family participated in study previously
* Caregiver's child was initially admitted to a unit besides the TCU
* Caregiver's child is NOT part of a service for which pediatric residents or advance practice providers provide care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of protocol implementation | 6 months after first meeting of protocol committee
  Feasibility of developing and implementing a social needs screening and intervention - measured dichotomously (yes/no) whether the protocol was developed and implemented within 6 months
Acceptability of social needs screening | Up to 6 months post baseline data collection
  Caregiver acceptability will be assessed using baseline surveys administered during inpatient recruitment in the pre-/ and post-protocol implementation periods. Care team member acceptability will be assessed using surveys administered after protocol implementation - Likert scale derived from De Marchis et al.'s 2019 paper: Do you think it is appropriate to be asked questions about your social and economic needs during your child's hospitalization? a) Very appropriate b) Somewhat appropriate c) Neither appropriate nor inappropriate d) Somewhat inappropriate e) Very inappropriate

SECONDARY OUTCOMES:
Recruitment rate | Up to 12 months after first meeting of protocol committee
  Proportion of caregivers recruited out of 50
Retention retention rate | Up to 15 months after first meeting of protocol committee
  Proportion of caregivers recruited that answer a post-hospitalization survey
Social needs screening rate | Up to 12 months after first meeting of protocol committee
  Proportion of families screened for social needs in the hospital
Caregiver-care team relationships | Up to 15 months after first meeting of protocol committee
  Assessments of the experience of caregivers with healthcare staff - Likert scale derived from De Marchis et al. 2019's paper: : How much do you trust your health care provider(s) at this hospital? 1 (not at all) through 10 (completely)
Family social needs | Up to 15 months after first meeting of protocol committee
  Depending on what social needs the inpatient unit decides to screen for (e.g., food insecurity, transportation needs), the investigators will measure the rates of those needs at the time of recruitment and then again 3 months post-discharge - dichotomous (i.e., presence or absence of food insecurity; presence or absence of transportation needs)
Child health status | Up to 15 months after first meeting of protocol committee
  Caregiver-endorsed measures of child health - Likert scale as derived from Gottlieb et al.'s 2020 paper: In general, would you say your child's health is: Excellent, very good, good, fair, poor
Rehospitalization rate | Up to 15 months after first meeting of protocol committee
  Proportion of children being readmitted within 3 months after discharge as reported by the caregiver
Post-hospitalization emergency department visit rate | Up to 15 months after first meeting of protocol committee
  Proportion of children being having an emergency department visit within 3 months after discharge as reported by the caregiver
Missed follow-up visit rate | Up to 15 months after first meeting of protocol committee
  Proportion of children missing a follow-up visit within 3 months after discharge as reported by the caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Pantell, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- Benioff Children's Hospital - San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot trial to examine the feasibility and acceptability of conducting a larger trial: 1) the study sample will be small and the investigators do not want to increase the risk of participant identification; 2) the pilot will not be powered enough to answer research questions related to outcomes for which other researchers might want to examine the data.

REFERENCES:
- [Background] Gottlieb LM, Adler NE, Wing H, Velazquez D, Keeton V, Romero A, Hernandez M, Munoz Vera A, Urrutia Caceres E, Arevalo C, Herrera P, Bernal Suarez M, Hessler D. Effects of In-Person Assistance vs Personalized Written Resources About Social Services on Household Social Risks and Child and Caregiver Health: A Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e200701. doi: 10.1001/jamanetworkopen.2020.0701. PMID 32154888
- [Background] De Marchis EH, Hessler D, Fichtenberg C, Adler N, Byhoff E, Cohen AJ, Doran KM, Ettinger de Cuba S, Fleegler EW, Lewis CC, Lindau ST, Tung EL, Huebschmann AG, Prather AA, Raven M, Gavin N, Jepson S, Johnson W, Ochoa E Jr, Olson AL, Sandel M, Sheward RS, Gottlieb LM. Part I: A Quantitative Study of Social Risk Screening Acceptability in Patients and Caregivers. Am J Prev Med. 2019 Dec;57(6 Suppl 1):S25-S37. doi: 10.1016/j.amepre.2019.07.010. PMID 31753277
- [Background] Gottlieb LM, Hessler D, Long D, Laves E, Burns AR, Amaya A, Sweeney P, Schudel C, Adler NE. Effects of Social Needs Screening and In-Person Service Navigation on Child Health: A Randomized Clinical Trial. JAMA Pediatr. 2016 Nov 7;170(11):e162521. doi: 10.1001/jamapediatrics.2016.2521. Epub 2016 Nov 7. PMID 27599265
- [Background] University of California, San Francisco Learning & Organization Development Employee Engagement. "Gallup Engagement Survey." Last accessed online on 10/8/2020: https://devlearning.ucsf.edu/gallup
- [Background] Gold R, Bunce A, Cottrell E, Marino M, Middendorf M, Cowburn S, Wright D, Mossman N, Dambrun K, Powell BJ, Gruss I, Gottlieb L, Dearing M, Scott J, Yosuf N, Krancari M. Study protocol: a pragmatic, stepped-wedge trial of tailored support for implementing social determinants of health documentation/action in community health centers, with realist evaluation. Implement Sci. 2019 Jan 28;14(1):9. doi: 10.1186/s13012-019-0855-9. PMID 30691480
- [Background] Schickedanz A, Hamity C, Rogers A, Sharp AL, Jackson A. Clinician Experiences and Attitudes Regarding Screening for Social Determinants of Health in a Large Integrated Health System. Med Care. 2019 Jun;57 Suppl 6 Suppl 2(Suppl 6 2):S197-S201. doi: 10.1097/MLR.0000000000001051. PMID 31095061
- [Background] Pantell MS, Kaiser SV, Torres JM, Gottlieb LM, Adler NE. Associations Between Social Factor Documentation and Hospital Length of Stay and Readmission Among Children. Hosp Pediatr. 2020 Jan;10(1):12-19. doi: 10.1542/hpeds.2019-0123. PMID 31888952
- [Background] Glick AF, Tomopoulos S, Fierman AH, Trasande L. Disparities in Mortality and Morbidity in Pediatric Asthma Hospitalizations, 2007 to 2011. Acad Pediatr. 2016 Jul;16(5):430-437. doi: 10.1016/j.acap.2015.12.014. Epub 2016 Jan 6. PMID 26768727
- [Background] Kaiser SV, Bakel LA, Okumura MJ, Auerbach AD, Rosenthal J, Cabana MD. Risk Factors for Prolonged Length of Stay or Complications During Pediatric Respiratory Hospitalizations. Hosp Pediatr. 2015 Sep;5(9):461-73. doi: 10.1542/hpeds.2014-0246. PMID 26330245
- [Background] Boyle CA, Decoufle P, Yeargin-Allsopp M. Prevalence and health impact of developmental disabilities in US children. Pediatrics. 1994 Mar;93(3):399-403. PMID 7509480
- [Background] Dell SD, Parkin PC, Macarthur C. Childhood asthma admissions: determinants of short stay. Pediatr Allergy Immunol. 2001 Dec;12(6):327-30. doi: 10.1034/j.1399-3038.2001.0s079.x. PMID 11846870
- [Background] Carroll CL, Uygungil B, Zucker AR, Schramm CM. Identifying an at-risk population of children with recurrent near-fatal asthma exacerbations. J Asthma. 2010 May;47(4):460-4. doi: 10.3109/02770903.2010.481344. PMID 20528602
- [Background] Macy ML, Stanley RM, Sasson C, Gebremariam A, Davis MM. High turnover stays for pediatric asthma in the United States: analysis of the 2006 Kids' Inpatient Database. Med Care. 2010 Sep;48(9):827-33. doi: 10.1097/MLR.0b013e3181f2595e. PMID 20706158
- [Background] Lin HC, Kao S, Wen HC, Wu CS, Chung CL. Length of stay and costs for asthma patients by hospital characteristics--a five-year population-based analysis. J Asthma. 2005 Sep;42(7):537-42. doi: 10.1080/02770900500214783. PMID 16169785
- [Background] Srivastava R, Homer CJ. Length of stay for common pediatric conditions: teaching versus nonteaching hospitals. Pediatrics. 2003 Aug;112(2):278-81. doi: 10.1542/peds.112.2.278. PMID 12897273
- [Background] Alderwick H, Gottlieb LM. Meanings and Misunderstandings: A Social Determinants of Health Lexicon for Health Care Systems. Milbank Q. 2019 Jun;97(2):407-419. doi: 10.1111/1468-0009.12390. Epub 2019 May 8. PMID 31069864
- [Background] Beck AF, Cohen AJ, Colvin JD, Fichtenberg CM, Fleegler EW, Garg A, Gottlieb LM, Pantell MS, Sandel MT, Schickedanz A, Kahn RS. Perspectives from the Society for Pediatric Research: interventions targeting social needs in pediatric clinical care. Pediatr Res. 2018 Jul;84(1):10-21. doi: 10.1038/s41390-018-0012-1. Epub 2018 May 23. PMID 29795202